CLINICAL TRIAL: NCT05522231
Title: A Phase II/III Clinical Study to Evaluate the Efficacy and Safety of Fruquintinib in Combination With Sintilimab Versus Axitinib or Everolimus as Second-line Treatment for Locally Advanced or Metastatic Renal Cell Carcinoma (FRUSICA-2)
Brief Title: Efficacy and Safety of Fruquintinib in Combination With Sintilimab in Advanced Renal Cell Carcinoma (FRUSICA-2)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-013-00CH1
Record Dates: First submitted 2022-08-16; First posted 2022-08-30 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Advanced Renal Cell Carcinoma
MeSH Terms: interventions — HMPL-013; sintilimab; Axitinib; Everolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational arm (Experimental): fruquintinib, 5 mg, QD, PO, 2 weeks on/1 week off, 3 weeks/cycle; sintilimab, 200 mg, IV infusion, Q3W, 3 weeks/cycle.
  Interventions: Drug: fruquintinib+sintilimab
- Control arm (comparator) (Active Comparator): axitinib, 5 mg, twice daily (BID), PO, 3 weeks/cycle, dose escalation will be at the investigator 's discretion ;Everolimus, 10 mg, QD, PO, 3 weeks/cycle.
  Interventions: Drug: axitinib / everolimus
- Fruquintinib monotherapy factorial study (Other): fruquintinib, 5 mg, QD, PO, 3 weeks on/ 1 week off, 4 weeks/cycle.
  Interventions: Drug: fruquintinib

INTERVENTIONS:
Drug: fruquintinib+sintilimab — fruquintinib, 5 mg, QD, PO, 2 weeks on/1 week off, 3 weeks/cycle; sintilimab, 200 mg, IV infusion, Q3W, 3 weeks/cycle.
  Other Names: HMPL-013 + IBI308
  Arms: Investigational arm
Drug: axitinib / everolimus — axitinib, 5 mg, twice daily (BID), PO, 3 weeks/cycle, dose escalation will be at the investigator 's discretion based on clinical; everolimus, 10 mg, QD, PO, 3 weeks/cycle.
  Arms: Control arm (comparator)
Drug: fruquintinib — fruquintinib, 5 mg, QD, PO, 3 weeks on/ 1 week off, 4 weeks/cycle.
  Other Names: HMPL-013
  Arms: Fruquintinib monotherapy factorial study

SUMMARY:
The study consists of two parts, the first part is a randomized, open-label, active-controlled study to evaluate the efficacy and safety of fruquintinib in combination with sintilimab versus axitinib or everolimus monotherapy as second-line treatment for locally advanced or metastatic renal cell carcinoma. The second part is a fruquintinib monotherapy factorial cohort study to evaluate the efficacy and safety of fruquintinib monotherapy as for second-line treatment of locally advanced or metastatic renal cell carcinoma.

DETAILED DESCRIPTION:
The target populations for this study were patients with histologically or cytologically confirmed, locally advanced/ metastatic renal cell carcinoma who progressed during or after or intolerant to previous first-line VEGFR-TKI therapy.

A total of about 249-264 patients are planned to be enrolled in the study, among whom about 234 patients are planned to be enrolled in the first part. The patients who are successfully enrolled will be randomly assigned into the investigational arm or the control arm in a 1:1 ratio. The enrollment of part 2 will be started after that of part 1 is completed. About 15~30 patients are planned to be enrolled in the second part. The patients who are successfully enrolled will receive fruquintinib monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 (inclusive) years of age on the date when ICF was signed;
2. Histologically or cytologically confirmed renal clear cell carcinoma;
3. Patients with locally advanced/metastatic renal carcinoma;
4. Patients with renal carcinoma who progressed during or after or intolerant to previous first-line VEGFR-TKI therapy for advanced/metastatic disease;
5. At least 1 measurable lesion according to RECIST 1.1;
6. ECOG PS of 0 or 1;
7. Adequate organ function.

Exclusion Criteria:

1. Had previously received therapy targeting immune modulatory receptors or related pathways (including but not limited to therapy targeting PD-1, CTLA-4, IDO, PD-L1, LAG-3, TIGIT, IL-2R and GITR, etc, but excluding related cytokine therapy such as IL2), excluding patients who had received immunotherapy such as anti-PD- (L) 1 antibody in adjuvant/neoadjuvant therapy setting and did not progress within 6 months after discontinuation;
2. Receiving approved systemic anti-tumor therapy within 2 weeks prior to the first dose;
3. Toxicities caused by prior anti-tumor therapy before the first dose that did not recover to Grade 0 or 1 per the NCI CTCAE v5.0 or to the level specified in the enrollment criteria (excluding alopecia and peripheral neurotoxicity ≤ CTCAE Grade 2);
4. Immunosuppression medication within 4 weeks prior to randomization;
5. Patients with active autoimmune or inflammatory diseases;
6. Known central nervous system (CNS) metastasis;
7. History of pneumonitis requiring corticosteroid therapy, or history of or current interstitial lung disease, or current active pulmonary infection, etc.;
8. Toxicities caused by prior anti-tumor therapy before the first dose that did not recover to Grade 0 or 1 per the National Cancer Institute Common Terminology Criteria for Adverse events (NCI CTCAE) v5.0 or to the level specified in the enrollment criteria (excluding alopecia and peripheral neurotoxicities ≤CTCAE Grade 2 caused by platinum-based chemotherapy; thyroid dysfunction with stable disease control after symptomatic treatment);
9. Human Immunodeficiency Virus (HIV) Infection (HIV 1/2 Antibody positive);
10. Uncontrolled hypertension despite standard therapy;
11. Patient with evidence or history of haemorrhagic tendency within 2 months prior to the first dose, regardless of severity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) in Part I | Time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months.
  PFS per RECIST 1.1 by BIRC
Objective response rate (ORR) in Part II | Time from the date of first treatment administration until disease progression or the introduction of a new treatment, assessed up to 20 months.
  ORR per RECIST 1.1 by investigator

SECONDARY OUTCOMES:
PFS | Time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months.
  PFS per RECIST 1.1
Safety in Part I | Through study completion, assessed up to 20 months.
  Severity and Incidence of Adverse event (AEs) and findings in Laboratory test, vital signs, 12-lead Electrocardiogram (ECG), etc. in Part I
Quality of life in Part I | Through study completion, assessed up to 20 months.
  Quality of life questionnaire analysis in Part I
Safety in Part II | Through study completion, assessed up to 20 months.
  Severity and incidence of AEs and findings in such as Laboratory test, vital signs, 12-lead ECG, etc. in Part II.
Disease control rate (DCR) | Time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months.
  PFS per RECIST 1.1
ORR | Time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months.
  ORR per RECIST 1.1
Duration of response (DoR) | Time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months.
  DoR per RECIST 1.1
Time to Response (TTR) | Time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months.
  TTR per RECIST 1.1
OS | Time from date of randomization until the date of death from any cause, assessed up to 20 months.
  OS

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Principal Investigator — Fudan University; Zhi Song He, Principal Investigator — Peking University First Hospital
Locations (48):
- China (48):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - The First Affilated Hospital of Fujian Medical University, Fuzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Harbin Medical University Cancer Hospital, Ha’erbin
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Qilu Hospital of Shandong University, Jinan
  - Shandong Cancer Hospital & Institute, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Lanzhou University Second Hospital, Lanzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Guangxi Medical University Cancer Hospital, Nanning
  - Nantong Tumor Hospital, Nantong
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Renji Hospital,Shanghai Jiaotong University School of Medicine, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Liaoning Cancer Hospital & Institution, Shenyang
  - The First Hospital of China Medical University, Shenyang
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou medical university, Wenzhou
  - Tongji Hospital Tongji Medical College of HUST, Wuhan
  - Wuhan Union Hospital of China, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiaotong University (Xibei Hosiptal), Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Henan Cancer Hospital, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No